CLINICAL TRIAL: NCT04047966
Title: Study of the Fetal and Maternal Microbiota in Preganant Women With Fetal Defect Growth Nad Its Relationship With Inflammatory Biomarkers
Brief Title: Study of the Fetal and Maternal Microbiota in Preganant Women With Fetal Defect Growth
Acronym: BIOCIR
Status: Terminated | Type: Observational
Why Stopped: Due to the current pandemic situation, recruitment has been disrupted by the inability to recruit more patients
Sponsor: Universidad de Granada (Other)
Collaborators: Hospital Sant Joan de Deu (Other)
Responsible Party: Principal Investigator, Carolina Gómez Llorente, Principal Investigator, Universidad de Granada
Other Study IDs: UGranada
Record Dates: First submitted 2019-07-11; First posted 2019-08-07 (Actual); Last update posted 2020-11-05 (Actual); Status verified 2020-11

CONDITIONS: Intrauterine Growth Restriction
Keywords: Intrauterine Growth restriction; Gastrointestinal microbiome; Inflammatory biomarkers
MeSH Terms: conditions — Fetal Growth Retardation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — We will recruit fecal samples to obtain bacterial DNA for metagenomics analysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Fetal growth restriction: 63 fetuses with defects in fetal growth qith an estimated fetal weight below 10th percentile
- Control group: 63 control fetuses with an estimated fetal weight about the 10th percentile

SUMMARY:
It is an observational and prospective study that will include consecutively 63 controls (fetuses with estimated fetal weight above the 10th centile) and 63 fetuses with defects in fetal growth (estimated fetal weight below the 10th percentile) during the third trimester (32-26 weeks) with gestational age at birth equal or over 37 weeks. Investigators will collect: (1) Obstetric and nutritional questionnaires, (2) maternal samples between 32-36 weeks (feces), (3) intrapartum samples (maternal blood, cord blood and placenta) and (4) postpartum samples (meconic and newborn feces at 6 weeks of life)

DETAILED DESCRIPTION:
It is an observational and prospective study to determine the influence of the gastrointestinal microbiome on the intrauterine growth restriction (IUGR). For this purpose, investigators are planning to recruit 63 women with a diagnoses of IUGR and 63 pregnant women with a normal intrauterine growth.

Samples will be taken during third trimester (fecal and blood maternal sample), intrapartum (maternal blood, umbilical cord blood and placenta tissue sample) and post partum samples (meconic and newborn fecal samples at 6 weeks of life).

Also, obstetric and nutritional information will be registered by means of specific questionnaires.

Fecal samples will be use to study the gastrointestinal microbiome by Next Generation Sequencing techniques, whereas inflammatory biomarkers will be determine in plasma samples.

ELIGIBILITY:
Inclusion Criteria:

* Intrauterine Growth restriction (32-36 weeks)
* Vaginal delivery
* Delivery at 37 weeks

Exclusion Criteria:

* Alcohol, tabacco or other drugs consumption during pregnancy
* Antibiotic use before recruitment (3 months) or during pregnancy until delivery
* Gestational diabetes
* Fetuses anormalities

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Study Population: 63 controls (fetuses with estimated fetal weight above the 10th centile) and 63 fetuses with defects in fetal growth (estimated fetal weight below the 10th percentile) during the third trimester (32-26 weeks) with gestational age at birth equal or over 37 weeks.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2018-03-02 (Actual); Primary Completion 2020-10-31 (Actual); Study Completion 2020-10-31 (Actual)

PRIMARY OUTCOMES:
Gastrointestinal microbiome composition (16S RNA amplicon sequencing) | From May to July 2020
  To determine the main gastrointestinal microbiota composition, by 16S RNA amplicon sequencing, in fecal samples of pregnant women and their newborn (meconic)

SECONDARY OUTCOMES:
Plasma levels of inflammatoy biomarkers | From May to July 2020
  To determine plasma inflammatory biomarkers levels (LPS, LBP, IL6, 8, 10, 13,15 IFN-gamma, VEGF) in pregnant woman by inmunoassay determination

CONTACTS AND LOCATIONS:
Overall Officials: Carolina Gomez Llorente, PhD, Principal Investigator — Universidad de Granada
Locations (1):
- Obstetrics and Gynecology, Hospital Sant Joan de Déu, Barcelona, Spain